CLINICAL TRIAL: NCT03409224
Title: Differences in Immunologic Response to Cryoablation Versus Radiofrequency Ablation in the Treatment of Renal Cell Carcinoma
Status: Terminated | Type: Observational
Why Stopped: not enough participants
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-6735
Record Dates: First submitted 2016-12-12; First posted 2018-01-24 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Immune Response to 3 Approaches

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Small cancer tissue samples were collected post ablation therapy.

GROUPS / COHORTS (1):
- Adults 18-99: Adults who are undergoing cryoablation

SUMMARY:
The purpose of this study is to compare changes in the body's self-defense (immune response) after two different treatments for small kidney tumors: 1) Cryoablation (freezing) therapy in which the tumor and a margin of normal kidney tissue are frozen and thawed twice with a needle probe and 2) radiofrequency ablation (RFA) in which radiofrequency energy delivered through a needle probe is used to heat tissue and thereby destroy a tumor.

ELIGIBILITY:
Inclusion Criteria:

* You are eligible to participate in this study if you are an adult (older than 18 years)
* Diagnosed with renal cell cancer 1-3 centimeters in size on the CT scan.

Exclusion Criteria:

* You are not eligible to participate in this study if you are immune compromised (chemotherapy,corticosteroid use, HIV [as documented in your medical record], etc.)
* Have an autoimmune disorders (Rheumatoid arthritis, Crohn's disease, etc)
* Have a tumor larger than 4 cm
* Are pregnant.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients that undergo one of the three treatments for Renal Masses:
  * Cryoablation
  * Partial Nephrectomy
  * Radiofrequency
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2003-01; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Immune Response to Cryoablation, RFA and Laparoscopic Partial Nephrectomy | 4 years
  The number of leukocytes found in the tissues cryoablation, radiofrequency ablation, or laparoscopic partial nephrectomy (control)